CLINICAL TRIAL: NCT02519608
Title: Comparison Between Ticagrelor and Clopidogrel Effect on Endothelial, Platelet and Inflammation Parameters in Patients With Stable Coronary Artery Disease and Chronic Obstructive Pulmonary Disease Undergoing PCI
Brief Title: ComparisoN of ticAgrelor vs. Clopidogrel in endoTHeliAl Function of COPD patieNts
Acronym: NATHAN-NEVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Assistant Professor and Interventional Cardiologist, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150497
Record Dates: First submitted 2015-07-31; First posted 2015-08-11 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; stable coronary artery disease; ticagrelor; clopidogrel; endothelial function; inflammation; platelet reactivity
MeSH Terms: conditions — Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Aspirin; Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin 100 mg + Clopidogrel 75 mg (Active Comparator): dual antiplatelet therapy as suggested by guidelines with aspirin 100 mg and clopidogrel 75 mg daily
  Interventions: Drug: Aspirin 100 mg; Drug: Clopidogrel
- Aspirin 100 mg + Ticagrelor 90 mg x2 (Experimental): dual antiplatelet therapy with aspirin 100 mg and ticagrelor 90 mg x 2 daily
  Interventions: Drug: Aspirin 100 mg; Drug: Ticagrelor

INTERVENTIONS:
Drug: Aspirin 100 mg — Patients with COPD and SCAD undergoing PCI and stent implantation will receive aspirin
  Other Names: baseline background treatment
Drug: Ticagrelor — Patients with COPD and SCAD undergoing PCI and stent implantation will receive according randomization aspirin + ticagrelor (loading dose 180 mg + maintenance 90 mg x2)
  Other Names: new hypothesis group
  Arms: Aspirin 100 mg + Ticagrelor 90 mg x2
Drug: Clopidogrel — Patients with COPD and SCAD undergoing PCI and stent implantation will receive according randomization aspirin + clopidogrel (loading dose 600 mg + maintenance 75 mg)
  Other Names: gold standard P2Y12 treatment
  Arms: Aspirin 100 mg + Clopidogrel 75 mg

SUMMARY:
This is an investigator-initiated, prospective, single-centre, randomised, phase II, open-label study, testing the superiority of ticagrelor, as compared to clopidogrel, in modulating on-P2Y12 treatment platelet reactivity, endothelial dysfunction and inflammation in chronic obstructive pulmonary disease (COPD) patients receiving scheduled percutaneous coronary intervention (PCI) for stable coronary artery disease. Subjects that meet the inclusion criteria and have provided informed consent will be randomly assigned in a 1:1 fashion to one of the two dual antiplatelet therapy (DAPT) regimen: aspirin + clopidogrel (standard of care) vs. aspirin + ticagrelor (experimental arm).

DAPT with aspirin and clopidogrel for at least 6 months (preferably 12 months) is the current gold-standard for patients receiving PCI and drug eluting stent implantation for SCAD. No data supports a different strategy and/or approach in COPD patients undergoing PCI. Ticagrelor, a new P2Y12 inhibitor, showed a significantly higher platelet inhibition as compared to clopidogrel. Recently, ticagrelor administration has been associated with a positive effect on endothelial function and a modulation of proinflammatory signalling. These actions are mediated by a significant influence of adenosine uptake. Higher platelet reactivity, chronic inflammatory response, heightened endothelial dysfunction characterized COPD patients with concomitant coronary artery disease (CAD). The investigators speculated that COPD patients undergoing PCI for stable CAD (SCAD) had a risk profile similar to that of acute coronary syndromes (ACS) patients. Accordingly, COPD patients undergoing PCI for SCAD may obtain a stronger benefit by ticagrelor as compared to clopidogrel. The aim of this study is to evaluate whether ticagrelor, is superior to clopidogrel, in reducing endothelial dysfunction , platelet reactivity (PR) and inflammation profile of patients with stable CAD and COPD. Ticagrelor will be administered according PLATO trial and international guidelines (180 mg as loading dose, 90 mg x 2 daily as maintenance dose). As suggested by international guidelines, the control group will be patients with current gold standard treatment for SCAD treated with PCI (aspirin + clopidogrel 75 mg daily). The evaluation of endothelial dysfunction, PR and inflammation profile will be repeated after 30 days and will be compared to baseline values.

DETAILED DESCRIPTION:
* Epidemiology Ischemic heart disease (IHD) and chronic obstructive pulmonary disease (COPD) are respectively the first and fourth cause of death in industrialized countries accounting for 10-15% of total disability adjusted life year (DALY). COPD is common in IHD patients, ranging from 5% to 18%, with a high prevalence of under diagnosis (until 87%). At the same time, one third of COPD patients' deaths are attributable to IHD and for every 10% decrease in forced expiratory volume in one second (FEV1), cardiovascular (CV) mortality rises by 28%.
* Prognostic implication of IHD-COPD comorbidity Presence of concomitant COPD and IHD has a negative impact on quality of life, disease progression and short and long-term outcome. After coronary revascularization patients with COPD are at higher risk of recurrent myocardial infarction (MI), heart failure (HF) and bleeding complications if compared to patients without COPD. Consequently, COPD is an independent predictor of mortality in MI patients (HR 1.4; 95%CI 1.2-1.6). In a retrospective study, including patients undergoing percutaneous coronary intervention (PCI) with a 4-years follow-up, COPD was an independent risk factor for all-cause mortality (odds ratio [OR], 1.79; 95%CI, 1.63-1.96), cardiac mortality (OR 1.57; 95%CI, 1.35-1.81), and occurrence of MI (OR 1.3; 95%CI, 1.14-1.47). Another prospective study on 5000 consecutive patients with coronary artery disease (CAD) evaluated the in-hospital period after PCI. Patients with COPD experienced a significantly higher incidence of angina (p<0.001), arrhythmias (p<0.001), composite major adverse cardiac events (p<0.001) and longer hospital stay (p<0.001) than patients without COPD. The analysis of Charlson index for stable CAD patients confirmed that the presence of COPD was strongly related with long-term survival.
* Inflammation, hypoxia and endothelial dysfunction COPD is characterized by a state of chronic inflammation of airways and vessels. Interleukin-6, C-reactive protein (CRP) and fibrinogen are often elevated in COPD and they facilitate both endothelial dysfunction and atherosclerosis progression. Fibrinogen induces plaque growing, stimulates platelets and white blood cells adhesion to vessels wall and promotes muscle cell proliferation and migration. Higher plasma levels of fibrinogen are directly related to a higher risk of acute coronary syndrome (ACS). CRP facilitates the production of interleukins and promotes the inflammatory state. Chronic hypoxia, contributing to endothelial dysfunction and increasing arterial stiffness, triggers, in vulnerable subjects, the growth and destabilization of atherosclerotic plaques.
* Platelet reactivity Heightened on-treatment PR is a well-known determinant of poor prognosis in PCI patients and it is significantly higher in COPD patients. In COPD patients, platelets' count tents to be higher, and thrombocytosis is associated with increased 1-year mortality (OR 1.53; 95% CI 1.03 to 2.29, p=0.03).
* Ticagrelor Ticagrelor is a direct-acting reversely binding inhibitor of P2Y12 platelets' receptor. Dual antiplatelet therapy (DAPT) with aspirin plus ticagrelor, as compared to aspirin plus clopidogrel, significantly reduces the rate of CV death, myocardial infarction, and/or stroke. Accordingly, DAPT with ticagrelor is guideline's recommended treatment (class I) in patients with ACS. On the contrary, DAPT with ticagrelor in stable CAD patients is not recommended. Dyspnea is a well-established ticagrelor potential side effect and it could be related to circulating increased adenosine levels after ticagrelor administration. A recent study by Alexopoulos et al. reported that COPD is a major determinant of poor/absent prescription of ticagrelor. Of note, Butler et al. demonstrated that ticagrelor administration does not alter pulmonary function at rest and during exercise in patients with COPD. Furthermore, ticagrelor-induced higher adenosine concentrations are considered the main mechanism of its "pleiotropic" effects (such as prevention of ADP-induced contraction of vascular smooth muscle cells, improvement of peripheral endothelial function and increase of endothelial nitric oxide synthase phosphorylation, reduction of pro-inflammatory thrombin-induced cytokines and chemokine's production during inflammation and coagulation activation).
* Research hypothesis and Rationale for conducting this study:

Many studies show that patients with COPD undergoing PCI and stent implantation are at higher risk of adverse events (death, MI and stent thrombosis, ST). This is true both for patients with ACS and stable coronary artery disease (SCAD). Many factors may explain this finding. First, COPD patients have a higher on-treatment (both aspirin and clopidogrel) platelet reactivity (PR). Second, inflammation profile is significantly enhanced in COPD, contributing to higher PR and endothelial dysfunction. Third, endothelial dysfunction due to hypoxia, abnormal shear stress and inflammation is common in COPD and may explain the increase of acute events after stent implantation. Patients receiving PCI and stent implantation must be treated with DAPT to minimize the risk of ST and recurrent MI. According current guidelines, DAPT should be started as soon as possible in patients with ACS and at the timing of PCI in patients with SCAD. Current guidelines recommended the association of aspirin and newer P2Y12 inhibitors (ticagrelor or prasugrel) for ACS patients, whereas aspirin and clopidogrel for SCAD patients. No data supports a different strategy and/or approach in COPD patients undergoing PCI. Ticagrelor, a new P2Y12 inhibitor, showed a significantly higher platelet inhibition as compared to clopidogrel. Recently, ticagrelor administration has been associated with a positive effect on endothelial function and a modulation of proinflammatory signalling. These actions are mediated by a significant influence of adenosine uptake. These findings support a possible positive effect of ticagrelor in COPD patients undergoing PCI for SCAD. Due to their comorbidity, COPD patients undergoing PCI for SCAD may be considered similar to ACS patients (higher platelet reactivity, chronic inflammatory response, heightened endothelial dysfunction). Accordingly, COPD patients undergoing PCI for SCAD may obtain a stronger benefit by ticagrelor when compared to clopidogrel. The aim of this study is to evaluate whether ticagrelor is superior to clopidogrel in reducing endothelial dysfunction, PR and inflammation profile of patients with stable CAD and COPD.

ELIGIBILITY:
Type of Patients Subjects either male or female eligible for PCI and undergoing drug eluting stent implantation who have meet all inclusion criteria and did not meet any of the exclusion criteria.

Inclusion Criteria:

For inclusion in the study subjects should fulfill the following criteria:

1. Age ≥18 years;
2. Ability to provide informed written consent and to participate in the 6-months follow-up period;
3. Diagnosis of SCAD requiring coronary artery angiography
4. COPD diagnosis confirmed by spirometry in stable phase and after medical treatment from at least 3 months.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Patients hospitalized with diagnosis of acute coronary syndrome
2. Previous chronic use of P2Y12 inhibitors
3. Known intolerance to aspirin and/or P2Y12 inhibitors
4. Absence of significant variation in guideline driven medical treatment in the last 15 days
5. History of intracranial haemorrhage
6. Known intake of a strong CYP3A4 inhibitor (e.g. ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir),
7. Known pregnancy, breast-feeding, or intend to become pregnant during the study period
8. Planned surgery, including CABG as a staged procedure (hybrid) within 6 months;
9. Known moderate to severe hepatic impairment (alanine-aminotransferase ≥ 3 x ULN);
10. Need for chronic oral anti-coagulation therapy;
11. Active major bleeding or major surgery within the last 30 days;
12. Known stroke (any type) within the last 30 days;
13. Currently participating in another trial before reaching primary endpoint;
14. Thrombocytopenia;
15. Increased risk of bradycardia;
16. Known other inflammatory chronic disorders;
17. Known or suspected malignancy
18. Other concomitant pulmonary diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
apoptosis rate in HUVEC | 1 month
  reduction of the rate of apoptosis in human umbilical vein endothelial cells (HUVEC) incubated with serum from patients enrolled in the study.

SECONDARY OUTCOMES:
on-treatment platelet reactivity | 1 month
  reduction of platelet reactivity (PR) as measured by P2Y12 and Aspirin VerifyNow System.
NO intracellular levels | 1 month
  modulation of intracellular levels of nitric oxid (NO) in HUVECs treated with serum from patients enrolled in the study
ROS production | 1 month
  reduction of intracellular levels of reactive oxygen species (ROS) in peripheral blood mononuclear cells (PBMCs) isolated from patients enrolled in the study
inflammation markers levels | 1 month
  reduction of values from baseline to 1 month of the most important inflammation cytokines associated with COPD (hs-PCR, fibrinogen, IL-6, IL-1Ra, TNF-alpha)
ischemic adverse events | 1 month
  Cumulative incidence of ischemic adverse events (death, myocardial infarction, stent thrombosis).
bleeding adverse events | 1 month
  Composite BARC 2-3-5 bleeding according to BARC definition
quality of life | 1 month
  Quality of life related to respiratory symptoms (COPD assessment test)

OTHER OUTCOMES:
apoptosis rate in HUVEC | time between LD and end of PCI, expected average of 5 hours
  rate of apoptosis in human umbilical vein endothelial cells (HUVEC) incubated with serum from patients enrolled in the study.
on-treatment platelet reactivity | time between LD and end of PCI, expected average of 5 hours
  reduction of platelet reactivity (PR) as measured by P2Y12 and Aspirin VerifyNow System.
NO intracellular levels | time between LD and end of PCI, expected average of 5 hours
  modulation of intracellular levels of nitric oxid (NO) in HUVECs treated with serum from patients enrolled in the study
inflammation markers levels | time between LD and end of PCI, expected average of 5 hours
  reduction of values from baseline to 1 month of the most important inflammation cytokines associated with COPD (hs-PCR, fibrinogen, IL-6, IL-1Ra, TNF-alpha)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

REFERENCES:
- [Result] Campo G, Vieceli Dalla Sega F, Pavasini R, Aquila G, Gallo F, Fortini F, Tonet E, Cimaglia P, Del Franco A, Pestelli G, Pecoraro A, Contoli M, Balla C, Biscaglia S, Rizzo P, Ferrari R. Biological effects of ticagrelor over clopidogrel in patients with stable coronary artery disease and chronic obstructive pulmonary disease. Thromb Haemost. 2017 Mar 23;117(6):1208-1216. doi: 10.1160/TH16-12-0973. Epub 2017 Mar 23. PMID 28331925